CLINICAL TRIAL: NCT06940479
Title: Genicular Artery Embolization for Knee Osteoarthritis: Evaluation of the Correlation Between Subjective Symptom Response and Objective Measures of Inflammation
Brief Title: Evaluating Changes in Synovial Fluid Before and After GAE for Knee Osteoarthritis
Acronym: GAE-KOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-1048
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GAE procedure (Other): Participants undergoing the GAE procedure will have synovial fluid sampling, performance-based measures and contrast-enhanced MRI before and after the procedure.
  Interventions: Procedure: GAE procedure

INTERVENTIONS:
Procedure: GAE procedure — Genicular artery embolization

SUMMARY:
The goal of this clinical trial is to learn if genicular artery embolization (GAE) can improve knee pain and decrease inflammation in adults with knee osteoarthritis. The main question it aims to answer is:

- Does the GAE procedure improve knee pain and decrease inflammation?

Researchers will compare synovial fluid samples taken from the knee before and after the procedure.

Participants will:

* Have a contrast enhanced MRI before and after the procedure
* Complete performance-based measures before and after the procedure
* Complete questionnaires before and after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planned to undergo genicular artery embolization to treat knee osteoarthritis.
* Osteoarthritis on knee radiograph (Kellgren-Lawrence score 1-3) within the last 6 months
* Persistent moderate to severe knee pain (visual analog scale [VAS] >3) for at least 6 months
* Pain refractory or intolerant to conservative therapies (e.g. analgesia, exercise, weight-loss, joint injections, physical therapy)
* BMI < 35 kg / m2
* Stated willingness to comply with study procedures and availability for the duration of the study

Exclusion Criteria:

* Coagulation disturbances not normalized by medical treatment (INR >1.8 and platelets <50 x 10^9/L)
* Receiving medications for anticoagulation which cannot safely be held for the procedure (e.g ASA for 5 days, Lovenox for 24 hours, Eliquis for 4-6 days depending on creatinine clearance
* Allergy to iodinated contrast agents not responsive to steroid premedication regimen
* Active knee joint infection
* Acute knee injury with surgical indication (MRI evidence of acute fracture or ligamentous injury of the knee)
* Prior total or partial knee replacement in the subject knee
* Intra-articular steroid injection within 2 months
* Untreated lower extremity vascular arterial disease
* Untreated venous insufficiency
* Presence of medical condition with life expectancy less than 6 months
* Patients who have undergone previous lower extremity embolization
* Patients with renal insufficiency based on an estimated GFR<45 ml/min who are not already on hemodialysis
* Patients who are pregnant or intend to become pregnant within 6 months of the procedure
* American Society of Anesthesiologists classification > 3
* Less than 3 mm of synovial fluid in the lateral suprapatellar recess on MRI or US

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Measure changes in KOOS score and synovial fluid biomarkers | 3 months after GAE procedure
  To estimate the correlation between objective changes in synovial fluid biomarkers (IL-6, VEGF and MCP-1) and changes in subjective symptomatic response (KOOS) 3 months after treatment of knee osteoarthritis with GAE.
  KOOS is a validated knee osteoarthritis scoring system that involves five subscales: pain (9 questions), symptoms (7 questions), activities of daily living (17 questions), sport/recreation (5 questions), knee-related quality of life (4 questions).
  Trials demonstrate maximum symptomatic response to GAE at 3 months, and sustained improvement for at least 1-2 years. Improvement in KOOS reflects symptomatic response to treatment. This will determine whether changes in the local inflammatory environment in the knee synovium correlate with symptomatic response to GAE. This would also help elucidate whether the mechanism of action of GAE is likely attributable to inflammation.

SECONDARY OUTCOMES:
Measure changes in synovial enhancement with contrast-enhanced MRI according to WORMS synovitis scores | 3 months after GAE procedure
  The WORMS scoring system is a semi-quantitative assessment of 14 features found on knee MRI. The WORMS synovitis subscale is scored based on the distension of the joint capsule and is graded from 0 to 3 in terms of the estimated maximal distention of the synovial cavity with 0=normal, grade 1=<33% of maximum potential distention grade 2=33%-66% of maximum potential distention and grade 3=>66% of maximum potential distention
  WORMS will be used to determine changes in synovial fluid biomarkers pre-treatment and 3 months after treatment of knee osteoarthritis with GAE.
Measure changes in synovial enhancement with contrast-enhanced MRI according to MOST grading system | 3 months after GAE procedure
  The MRI will also be evaluated using the Multicenter Osteoarthritis Study grading system for synovitis.
  The Multicenter Osteoarthritis Study (MOST) grading system for knee synovitis is an alternative to the WORMS synovitis score and incorporates a larger range of grading. The higher the score, the worse the synovial inflammation. The scoring ranges from 0-13, with 0-4 for normal or equivocal synovitis, 5-8 for mild synovitis, 9-12 for moderate synovitis, and 13 or greater for severe synovitis.
Measure changes in VAS scores | 12 months after procedure
  Patients will be given VAS questionnaires to give subjective responses to changes in pain levels and its effect on activities of daily living.
  VAS is calculated by scoring pain level between 0-100. This is asked verbally "How would you rate your pain in the affected knee?"
  These questionnaires will be given at time points: screening, 1 month after GAE, 3 months, 6 months and 12 months.
Measure changes in KOOS scores | 12 months after procedure
  The Knee Injury and Osteoarthritis Outcome Score involves five subscales: pain (9 questions), symptoms (7 questions), activities of daily living (17 questions), sport/recreation (5 questions), knee-related quality of life (4 questions).
  Patients will be given KOOS questionnaires to give subjective responses to changes in pain levels and its effect on activities of daily living.
  These questionnaires will be given at time points: screening, 1 month after GAE, 3 months, 6 months and 12 months.
Estimate correlation between objective measures to symptomatic response | 3 months after GAE procedure
  To estimate the correlation between objective measures of knee pain or inflammation (performance-based measures, contrast-enhanced MRI synovitis scores) to symptomatic response (KOOS) 3 months after treatment of knee osteoarthritis with GAE. This may provide additional assurance in the form of objective measures of response in a disease that is known to have a strong placebo effect.
Estimate correlation between changes in a larger set of synovial fluid biomarkers and changes in subjective scores | 3 months after GAE procedure
  To estimate the correlation between changes in a larger set of synovial fluid biomarkers (54markers across inflammation, chemotaxis, angiogenesis, and immune system regulation pathways) and changes in subjective scores (KOOS) 3 months after treatment. This will further develop the interrogation of which microenvironment pathways in the knee synovium correlate with symptomatic response to GAE.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Casadaban, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No